CLINICAL TRIAL: NCT00812825
Title: A Phase 1, Active and Placebo-Controlled, Multiple-Dose Escalation Trial Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-04171327 (Part 1), and a Single Dose Pharmacokinetic Assessment of a Tablet Formulation (Part 2) in Healthy Volunteers
Brief Title: A Phase 1 Multiple-Dose Escalation and Single Dose (Tablet) Study of PF-04171327 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A9391002
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Volunteers
Keywords: Safety Tolerability Pharmacokinetics/pharmacodynamics
MeSH Terms: interventions — fosdagrocorat; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- PF-04173127 (Experimental)
  Interventions: Drug: PF-04171327
- Prednisolone (Active Comparator)
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Solution Placebo (Sham Comparator)
  Interventions: Drug: Placebo Solution
- PF-04171327 Tablet (Experimental)
  Interventions: Drug: PF-04171327 Tablet

INTERVENTIONS:
Drug: PF-04171327 — PF-0417327 will be provided as an oral solution administered at doses of 1, 3, 10 and 30 mg. If an additional cohort is required, the dose selected will not exceed 100 mg. Solution will be administered once daily for 14 days.
  Arms: PF-04173127
Drug: Prednisolone — Oral doses of prednisolone (5, 10, and 20 mg) will be administered to the first three cohorts. The fourth cohort will receive between 1 and 20 mg to be determined after the third cohort completes dosing. If an additional cohort is required, the dose selected will not exceed 40 mg. Prednisolone tablets will be administered once daily for 14 days
  Arms: Prednisolone
Drug: Placebo — Tablets similar in appearance to prednisolone will be administered once daily for 14 days.
  Arms: Placebo
Drug: Placebo Solution — Placebo solution will be administered to those volunteers who are randomized to the placebo or prednisolone arms. This will be administered orally each day for 14 days.
  Arms: Solution Placebo
Drug: PF-04171327 Tablet — A single 10 mg dose of PF-04171327 tablet formulation will be administered orally to volunteers in Part 2 of this study.
  Arms: PF-04171327 Tablet

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics (how the drug effects certain target sites of activity in the body) of escalating doses of oral PF-04171327 in healthy volunteers for 14 days (Part 1). Part 2 will evaluate the pharmacokinetics of a single 10 mg dose of the PF-04171327 tablet in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 55 years, inclusive.
* Healthy females between 18 and 44 years, inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant disease;
* Post-menopausal women;
* History of intolerance or significant adverse effects with glucocorticoids. therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple doses of PF-04171327 | 14 days
Determination of pharmacokinetic parameters of PF-04171327 after multiple doses | 14 days
Assessment of the pharmacodynamic effects of PF-04171327 on chemical and metabolic biomarkers | 14 days
Evaluation of the pharmacokinetic parameters of a single 10 mg dose of PF-04171327 tablet | 1 day

SECONDARY OUTCOMES:
To characterize the pharmacodynamic effects of prednisolone | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9391002&StudyName=A%20Phase%201%20Multiple-Dose%20Escalation%20and%20Single%20Dose%20%28Tablet%29%20Study%20of%20PF-04171327%20in%20Healthy%20Volunteers